CLINICAL TRIAL: NCT02634931
Title: A Long-term, Single-arm, Open-label Trial of NPC-12G (Topical Formulation of Sirolimus) to Angiofibroma and Other Skin Lesions in Patients With Tuberous Sclerosis Complex
Brief Title: Long-term Trial of Topical Sirolimus to Angiofibroma in Patient With Tuberous Sclerosis Complex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-12G-2
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2015-12

CONDITIONS: Tuberous Sclerosis; Angiofibroma; Hypomelanotic Macule; Plaque
Keywords: Sirolimus; Skin lesions; TSC; Tuberous Sclerosis Complex; NPC-12G; Angiofibroma; Hypomelanotic Macule; Plaque
MeSH Terms: conditions — Tuberous Sclerosis; Angiofibroma; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPC-12G gel (Experimental): NPC-12G gel is containing 0.2% Sirolimus
  Interventions: Drug: NPC-12G gel

INTERVENTIONS:
Drug: NPC-12G gel — NPC-12G gel is administered topically twice a day for 52 weeks or longer

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of long-term treatment with NPC-12G gel (0.2% sirolimus gel) to angiofibroma and other skin lesions in patients with tuberous sclerosis complex in the open-label trial.

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is an autosomal dominant hereditary disease that causes benign tumors on the almost whole body (including skin, brain, kidney, lung and heart), behavior disorder as autism, mental retardation and neurologic symptom as epilepsy. Angiofibroma is a TSC-specific facial skin lesion, and hamartoma caused by increase of the component of skin connective tissues and blood vessels. Other skin lesions due to TSC are white macule (hypomelanotic macule), plaque, shagreen patch and ungual fibromas. Current therapeutic methods for angiofibroma are laser and surgical treatments, but there are problems as many relapses, deficiency of evidence, change of pigment, scar and risk of infection.

This is a multicenter and open-label trial. The trial consists of two phase. In the first trial phase for 52 weeks, the efficacy as well as the safety is evaluated. For the second trial phase the trial will be continued until the date of approval of NDA for NPC-12G. The safety is evaluated during the second trial phase, but not the efficacy. Patients who meet all entry criteria for the trial apply 0.2% NPC-12G gel twice a day. Patients will visit at 4 to 5-week intervals for the first 6 months of the first trial phase, and then 3 months intervals thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 3 years old or greater at the time of informed consent
2. Patients who are diagnosed as definite diagnosis according to diagnostic criteria for tuberous sclerosis complex (International Tuberous Sclerosis Complex Consensus Conference 2012)
3. Patients with skin lesions such as angiofibroma, white macules or plaque upper neck associated with tuberous sclerosis complex at the screening visit or the baseline visit
4. Patients or his/her guardian who agree to use the test drug (NPC-12G gel) or who want to participate in the trial again following participation in Phase III trial (NPC-12G-1)
5. Patient who are considered to be an appropriate patient to participate in the trial by investigator
6. Patients or his/her guardian who give a written informed consent in understanding and willingness after having received enough explanation of the test drug and the current trial plan

Exclusion Criteria:

1. Patients who have offered to withdraw from Phase III trial (NPC-12G-1) and have been discontinued
2. Patients who have not applied the test drug topically more than 25% of whole applications without appropriate reason for Phase III trial (NPC-12G-1)
3. Patients with clinical findings such as erosion, ulcer and eruption on or around the lesion of angiofibroma, which may affect assessment of safety or efficacy
4. Patients with a history of hypersensitivity to alcohol or allergy to sirolimus
5. Patients who have complications such as malignant tumor, infection, serious heart disease, hepatic function disorder, renal function disorder or blood disorders which severity are considered by investigator as grade 2 or more severe with reference to ''Concerning classification criteria for seriousness of adverse drug reactions of medical agents''
6. Patients who have complications such as diseases unsuitable for the trial participation, for examples, uncontrolled diabetes (fasting blood glucose level >140 mg/dL or postprandial blood glucose level > 200 mg/dL), dyslipidemia (cholesterol level > 300 mg/dL or > 7.75 mmol/L, triglycerides level > 300 mg/dL or > 3.42 mmol/L), etc.
7. Female patients who may be pregnancy or are lactating
8. Patients who cannot agree to take appropriate measures of contraception until completion of the trial or follow-up period after discontinuation from informed consent
9. Patients who have participated in other clinical trial other than Phase III trial (NPC-12G-1) and have taken a trial drug within 6 months before informed consent
10. Others, patients who are considered by the investigator as unsuitable for participation in the trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The discontinuation rate due to adverse events | 52 weeks and longer
  The first discontinuation in each patient due to adverse events is assessed.Completion of week 26 and 52 are cut-off points for interim-analyses by Kaplan-Meier method

SECONDARY OUTCOMES:
Adverse events and adverse events related to the test drug | 52 weeks and longer
  The number of discontinuation/ resume due to adverse events are evaluated. Completion of week 26 and 52 are cut-off points for interim-analyses
Adverse events related to the test drug leading to the discontinuation permanently | 52 weeks and longer
  The incidence of adverse events are evaluated. Completion of week 26 and 52 are cut-off points for interim-analyses
Serious adverse events and serious adverse events related to the test drug | 52 weeks and longer
  The incidence of serious adverse events are evaluated. Completion of week 26 and 52 are cut-off points for interim-analyses
Adverse events and adverse events related to the test drug leading to modification of dosage and administration | 52 weeks and longer
  The incidence of adverse events are evaluated. Completion of week 26 and 52 are cut-off points for interim-analyses
Significant adverse events and significant adverse events related to the test drug | 52 weeks and longer
  The incidence of significant adverse events such as local irritation are evaluated. Completion of week 26 and 52 are cut-off points for interim-analyses
Laboratory tests, vital signs | Baseline and every 3 months for laboratory tests, every scheduled visit for vital sign]
  Completion of week 26 and 52 are cut-off points for interim-analyses
Blood level of sirolimus | Baseline and every 3 months only for the first trial phase
  Whole blood level of sirolimus are measured any day time at baseline and every 3 months visit
Improvements in angiofibroma | Week 4, 8, 12, 26, 39 and 52
  Improvements comparing with baseline is assessed using photograph by the investigator and the central photo-judgement committee. Completion of week 26 is a cut-off point for interim-analysis.
Improvements in sizes of angiofibroma | Week 4, 8, 12, 26, 39 and 52
  Improvements comparing with baseline is assessed using photograph by the investigator and the central photo-judgement committee. Completion of week 26 is a cut-off point for interim-analysis.
Improvements in redness of angiofibroma | Week 4, 8, 12, 26, 39 and 52
  Improvements comparing with baseline is assessed using photograph by the investigator and the central photo-judgement committee. Completion of week 26 is a cut-off point for interim-analysis.
Improvements in white macule and plaque upper neck | Week 4, 8, 12, 26, 39 and 52
  Improvements comparing with baseline is assessed using photograph by the investigator and the central photo-judgement committee. Completion of week 26 is a cut-off point for interim-analysis.
The rate of patients evaluated ''improvement'' or more (improvement rate) in above the efficacy measures. | Week 4, 8, 12, 26, 39 and 52
  Completion of week 26 is a cut-off point for interim-analysis.
Change in total score of DLQI and CDLQI from baseline | Week 4, 8, 12, 26, 39 and 52
  DLQI for subjects 16 years old and greater, or CDLQI for children of less than 16 years old is assessed by patients. Completion of week 26 is a cut-off point for interim-analysis.
Degree of patient's satisfaction | Week 12, 26, 39 and 52
  Patient's satisfaction is assessed by patient. Completion of week 26 is a cut-off point for interim-analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mari Wataya-Kaneda,, MD, PhD, Principal Investigator — Department of Dermatology, Graduate School of Medicine, Osaka University
Locations (1):
- Graduate School of Medicine, Osaka University, Suita, Osaka, Japan

REFERENCES:
- [Derived] Wataya-Kaneda M, Nagai H, Ohno Y, Yokozeki H, Fujita Y, Niizeki H, Yoshida K, Ogai M, Yoshida Y, Asahina A, Fukai K, Tateishi C, Hamada I, Takahata T, Shimizu K, Shimasaki S, Murota H. Safety and Efficacy of the Sirolimus Gel for TSC Patients With Facial Skin Lesions in a Long-Term, Open-Label, Extension, Uncontrolled Clinical Trial. Dermatol Ther (Heidelb). 2020 Aug;10(4):635-650. doi: 10.1007/s13555-020-00387-7. Epub 2020 May 8. PMID 32385845